CLINICAL TRIAL: NCT02430740
Title: Multicentric Randomized Controlled Study to Determine a Tailored Strategy for Controlled Ovarian Stimulation in IVF Based on AMH, BMI and AFC
Brief Title: Tailored Ovarian Stimulation Based on BMI, AMH, AFC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Wyns, MD, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMH1
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Infertility
Keywords: Fertilization in Vitro; antagonist protocol; antral follicle count; Anti-Mullerian Hormone; Reproductive Techniques, Assisted
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — follitropin alfa; follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Other): standard care recFSH
  Interventions: Drug: recFSH
- study group (Experimental): modified dosage of recFSH for controlled ovarian stimulation based on AMH, BMI and AFC
  Interventions: Drug: recFSH

INTERVENTIONS:
Drug: recFSH
  Other Names: Gonal F; Puregon; Fostimon

SUMMARY:
The study objective is to develop a tailored based strategy for ovarian stimulation in IVF patients using AMH, BMI, antral follicle count (AFC).

300 patients will be randomized in 2 arms:

1. control group: standard care rec FSH.
2. study group: modified dose of Rec FSH based on AFC with a correction factor based on BMI and basal AMH level.

Primary endpoints: number of mature follicles and eggs collected at egg retrieval; amount of rec FSH used.

Secondary endpoints: fertilization rate; cleavage rate; clinical pregnancy rate; inhibin B and AMH levels during ovarian stimulation.

DETAILED DESCRIPTION:
The study objective is to develop a tailored based strategy for ovarian stimulation in IVF patients using AMH, BMI, AFC and inhibin B.

300 patients will be stimulated with rec FSH and an antagonist pituitary inhibition protocol, and randomized (at random computer generated numbers) in 2 arms:

1. control group: standard care recFSH based on age, basal FSH and AFC.
2. study group: modified dose of Rec FSH based on AFC with a correction factor based on BMI and basal AMH level.

FSH administration: 20IU per antral follicle (from 2-5mm) corrected as follows:

Correction factor for

AMH:

<1 pMol/L X4 1-6 pMol/L X2 7-18 pMol/L X1 >18 pMol/L X0.5 BMI 16.5-18.5 X0.75 18.5-25 X1 25-30 X1.25 30-35 X1.5 35-40 X2 Primary endpoints: number of mature follicles and eggs collected at egg retrieval; amount of rec FSH used.

Secondary endpoints: fertilization rate; cleavage rate; clinical pregnancy rate; inhibin B and AMH levels during ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* female infertile patients eligible for IVF treatment

Exclusion Criteria:

* polycystic ovaries
* untreated thyroid pathology
* hypogonadotropic hypogonadism
* untreaed hyperprolactinemia
* study drug hypersensitivity
* previous OHSS
* unilateral ovariectomy
* genital malformation
* BMI>40

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
number of mature follicles | 2 years
number of oocytes retrieved | 2 years
rec FSH dose used | 2 years

SECONDARY OUTCOMES:
fertilization rate | 2 years
cleavage rate | 2 years
clinical pregnancy rate | 2 years
AMH level during stimulation | 2 years
Inhibin B level during stimulation | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No